CLINICAL TRIAL: NCT01065415
Title: The Efficacy of Coregistered Whole-Body Magnetic Resonance Imaging/Positron Emission Tomography (MRI/PET) in the Staging of Non-Small-Cell Lung Cancer
Brief Title: Whole-Body Magnetic Resonance Imaging/Positron Emission Tomography (MRI/PET) in the Staging of Non-Small-Cell Lung Cancer (NSCLC)
Status: Completed | Type: Observational
Sponsor: Samsung Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2008-07-019
Record Dates: First submitted 2010-02-08; First posted 2010-02-09 (Estimated); Last update posted 2011-12-29 (Estimated); Status verified 2011-12

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Magnetic Resonance Imaging/Positron Emission Tomography; Whole body imaging; Non-small cell lung cancer; staging; Diagnostic accuracy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- control group: routine staging work-up with chest CT, PET/CT, and brain MRI
- study group: routine staging work-up plus whole body MRI for Coregistered MRI/PET

SUMMARY:
The accurate staging is an essential part for the treatment and prognosis of non-small-cell lung cancer (NSCLC). Whole body MR imaging proved to be effective in staging of NSCLC as much as PET/CT. And there were organs of strength for each modality in the detection of metastasis. Therefore, integrated approach using whole body MR and PET would be more beneficial for the accurate staging of lung cancer with improved diagnostic efficacies and reduced radiation exposure.

The aim of this project is to evaluate the diagnostic efficacy of side-by-side reading of whole-body magnetic resonance imaging/ positron emission tomography (MRI/PET) and to compare with that of whole-body magnetic resonance imaging (WB MRI) alone and that of integrated PET/CT in determining the stage of NSCLC.

Patients with pathologically-proven NSCLC will be prospectively enrolled, if they are considered as surgical candidates for the treatment of lung cancer through conventional methods of staging, i.e. history taking, physical examination, blood tests, bronchoscopy, and enhanced chest CT scans. PET/CT will be routinely performed for the staging of lung cancer in our institution. For the purpose of this study, whole body MRI will be performed for these patients within 3 days from the date of acquisition of PET/CT. The results of TNM staging from each modality will be collected prospectively and their efficacies can be calculated based on the reference standards. Reference standards of T and N staging will be surgically confirmed. And M staging can be confirmed by biopsy, other imaging modalities, or follow-up more than 6 months.

Diagnostic efficacies of coregistered MRI/PET can be evaluated with the comparison from the consecutive two-arm enrollment with random assignment of control group and study group as follows:

* control group: routine staging work-up with chest CT, PET/CT, and brain MRI
* study group: routine staging work-up plus whole body MRI for Coregistered MRI/PET

DETAILED DESCRIPTION:
Non-small cell lung cancer (NSCLC) accounts for 75 to 80% of all lung cancers, and is currently the leading cause of tumor-related deaths (1). Optimal lung cancer treatment relies on accurate disease staging, which is based on tumor size and extent, regional nodal involvement, and the presence of metastasis. Although thoracic CT has been considered the standard modality of choice for assessing intrathoracic spread of lung cancer (2), no consensus has been reached concerning metastasis evaluation. [18F]-fluorodeoxyglucose (FDG)-positron emission tomography (PET) was introduced and developed as an integrated modality for accurate nodal staging and for metastatic lesion detection in the whole body (WB) (3-9). Currently, integrated PET/CT, by providing both morphologic and metabolic features, appears to have achieved better efficacy in staging lung cancer than CT alone or PET alone (8, 10).

Whole body magnetic resonance imaging (WB MRI) has become feasible and enables fast scan throughout the body (11-13). This technique is based on a real-time gradient-echo imaging and sliding table platform (rolling table concept, which eliminates time-consuming repositioning of patients and surface coils). MRI scanners of the latest generation use high field MRI units of > 1.5 Tesla (T), and are reported to have upgraded capabilities in terms of temporal and spatial resolution due to improved signal-to-noise ratios (SNRs) under high magnetic-field strength conditions (14, 15).

Because both integrated PET/CT and WB MRI can provide WB imaging, both modalities are used for staging in patients with a malignant condition. According to a report (16), the diagnostic efficacy of PET/CT is superior to WB MRI for T and N staging and similar to WB MRI for detecting metastases. However, according to another study (17), WB MRI showed better sensitivity than PET/CT for detecting metastatic lesions. In these studies (16, 17), in which a 1.5T MR unit was used, the regional nodal or metastatic lesions were from various types of primary malignancies with a wide range of tumor stages.

Recently we published a paper regarding the diagnostic efficacy comparison for determining TNM stages of integrated PET/CT and 3T WB MRI in patients with an NSCLC (18). In this study, we found that both PET/CT and 3T whole body MRI appear to provide acceptable accuracy and comparable efficacy for non-small cell lung cancer staging, but in M stage determination, each modality has its own advantages. Namely, WB MRI is more useful for detecting brain and hepatic metastases, whereas PET/CT for lymph node and soft-tissue metastases. Therefore, we suggested whole body MR/PET should be the future imaging modality for NSCLC staging especially for M staging.

Although PET/CT scanners have quickly become established, development of MRI/PET has been slower, due to the additional challenge of developing dual-modality systems that avoid deleterious interactions caused by the high magnetic field environment of the MRI scanner and radiofrequency (RF) interference between the PET and MRI systems. At this moment, MRI/PET is still under development and is used only in small animal study (19). Thus, the purpose of this research is to provide clinical corroborating data to show how effective future MRI/PET will be in human use especially in patients with NSCLC by providing the efficiency of side-by-side reading of WB MRI/PET as compared to PET/CT.

ELIGIBILITY:
Inclusion Criteria:

* Patient with solitary pulmonary nodule under the suspicion of lung cancer
* Patients with NSCLC proved at pathologic examination will do PETCT as a routine staging work-up.

Exclusion Criteria:

* patients with contraindication for the MR scan such as metalic device or claustrophobia

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient under the suspicion of lung cancer or Patients with NSCLC proved at pathologic examination
Sampling Method: Probability Sample
Enrollment: 272 (Actual)
Dates: Start 2010-02; Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kyung Soo Lee, Prof., Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea

REFERENCES:
- [Derived] Yi CA, Lee KS, Lee HY, Kim S, Kwon OJ, Kim H, Choi JY, Kim BT, Hwang HS, Shim YM. Coregistered whole body magnetic resonance imaging-positron emission tomography (MRI-PET) versus PET-computed tomography plus brain MRI in staging resectable lung cancer: comparisons of clinical effectiveness in a randomized trial. Cancer. 2013 May 15;119(10):1784-91. doi: 10.1002/cncr.28000. Epub 2013 Feb 19. PMID 23423920